CLINICAL TRIAL: NCT02164344
Title: Effects of Probiotics on Microbial Translocation and Immune Activation Markers in HIV-positive Patients on Combined Antiretroviral Therapy and Non-virological Study of the Effects of Therapy
Brief Title: Effects of Probiotics on Microbial Translocation and Immune Activation Markers in HIV-positive Patients on Combined Antiretroviral Therapy
Acronym: PROBIO-HIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giancarlo Ceccarelli, MD, PhD, MSc, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DPHID-UniRoma03
Record Dates: First submitted 2014-06-11; First posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-03

CONDITIONS: HIV
Keywords: HIV; Gut; probiotics; immune activation
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Probiotics (Experimental): HIV-1 infected patients take daily dietary supplement with probiotics for at least 3 months
  Interventions: Dietary Supplement: probiotics

INTERVENTIONS:
Dietary Supplement: probiotics — probiotics (Streptococcus salivarius ssp. termophilus, Bifidobacterium breve, Bifidobacterium infantis, Bifidobacterium longum, Lactobacillus acidophilus, Lactobacillus plantarum, Lactobacillus casei, Lactobacillus delbrueckii ssp. bulgaricus and Streptococcus faecium)

SUMMARY:
Combined antiretroviral therapy (cART)-treated patients have increased mortality and morbidity compared to age-matched seronegative individuals. This increased mortality and morbidity has been associated to immune activation that persists also in patients under cART even with undetectable levels of HIV-RNA in blood. Indeed, HIV-infected patients, irrespective of cART treatment, show higher levels of activated T cells, inflammatory monocytes and proinflammatory cytokines than seronegative individuals. Several putative causes of this residual inflammation have been proposed and include ongoing HIV replication at low levels, the presence of coinfections such as cytomegalovirus, and microbial translocation.

None of these causes are mutually exclusive and understanding the degree to which of these three cause residual inflammation in cART-treated individuals will require novel therapeutic interventions aimed at alleviated each putative cause.

In this longitudinal study we aim:

1. to reduce microbial translocation induced inflammation in cART-treated individuals with supplementation of cART with the probiotics.
2. to investigate the potential benefits of 24 weeks of probiotics supplementation on immune function and on immune activation status

Indeed, the early stage of HIV infection is associated with dysbiosis of the GI tract microbiome with reducted levels of bifidobacteria and lactobacillus species with increased levels of potentially pathogenic proteobacteria species.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive patients
* HIV viral load < 50 copies/ml
* antiretroviral therapy from at least 2 years

Exclusion Criteria:

* intestinal diseases
* opportunistic diseases
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Delta of Cluster of Differentiation 4 (CD4)+/Cluster of Differentiation 38 (CD38)-/Human Leukocyte Antigen-D related (HLA-DR+) | 3 months
  Delta of CD4+/CD38-/HLA-DR+ in blood (T0-T1)

SECONDARY OUTCOMES:
Delta of Cluster of Differentiation 8 (CD8)+/CD38+/HLA-DR+ | 3 months
  Delta of CD8+/CD38-/HLA-DR+ in blood (T0-T1)
CD4 recovery (ΔCD4) | 3 months
  CD4 recovery (ΔCD4),in blood at T0 and T1

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Vullo, MD, Principal Investigator — University of Rome "Sapienza" (Italy)
Locations (2):
- Italy (2):
  - Department of Public Health and Infectious Diseases, University of Rome "Sapienza", Italy, Rome, RM
  - Department of Public Health and Infectious Diseases. University of Rome "Sapienza" (Italy), Rome

REFERENCES:
- [Derived] d'Ettorre G, Ceccarelli G, Giustini N, Serafino S, Calantone N, De Girolamo G, Bianchi L, Bellelli V, Ascoli-Bartoli T, Marcellini S, Turriziani O, Brenchley JM, Vullo V. Probiotics Reduce Inflammation in Antiretroviral Treated, HIV-Infected Individuals: Results of the "Probio-HIV" Clinical Trial. PLoS One. 2015 Sep 16;10(9):e0137200. doi: 10.1371/journal.pone.0137200. eCollection 2015. PMID 26376436